CLINICAL TRIAL: NCT06398860
Title: Effectiveness- and Cost Effectiveness of a Structured Method for Systematic and Integrated Occupational Safety and Health and Patient Safety Management Systems (SIOHPS) - A Pragmatic Stepped Wedge Cluster Randomised Controlled Trial
Brief Title: A Structured Method for Systematic and Integrated Occupational Safety and Health and Patient Safety Management Systems
Acronym: SIOHPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Collaborators: Uppsala University (Other); University of Gavle (Other); Karolinska Institutet (Other); Uppsala County Council, Sweden (Other Government); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Malin Lohela Karlsson, Associate professor, Region Västmanland
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-00404; 2022-00404 (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Sick Leave; Quality Of Care; Occupational Health; Safety Culture; Cost-effectiveness; Preventable Adverse Events; Patient Safety; Worker Health; Stress; Productivity Loss
Keywords: Work conditions; Patient safety; Health service; Intervention research; Stakeholder Participation; Co-production; Debrief; Safety huddle; Process evaluation
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: The study uses a stepped wedge cluster-controlled design with open cohort, where workplace acts as a cluster.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention-arm (Experimental): Cluster of 3-6 workplaces will start intervention at either baseline, 4 or 8 month from the start.
  Interventions: Procedure: SIOHPS
- Wait-list group (Experimental): Wait-listed group, will await intervention for either 4 or 8 months.
  Interventions: Procedure: Wait-list

INTERVENTIONS:
Procedure: SIOHPS — The intervention is comprised of several core components such as targeted education, daily team reflections and support for systematic management. First, a two hour education will be conducted for management, HCW involved in patient safety work, safety representatives and intervention facilitators. The second core component is a short daily team reflection conducted by HCW at the unit in connection to the end of work shifts. These are standardized to support identification of situations at work related to both Safety I and II perspective for both occupational health and patient safety as well as learning. The third component includes risk assessment, planning and implementation of appropriate measures, follow up and evaluation, based in information identified in the second component. The steps in this component targets the management and should be conducted in close collaboration with HCW involved in patient safety work and the safety representatives.
  Arms: Intervention-arm
Procedure: Wait-list — No intervention
  Arms: Wait-list group

SUMMARY:
The evidence unequivocally supports the association between work environment and patient safety. The negative impact of working conditions on both employee health and quality of care highlights the potential benefits of integrating these areas. It is therefore suggested that integrated systematic occupational health and patient safety management are crucial in managing the challenges faced by healthcare services today.

The project aims to assess the effectiveness and cost-effectiveness of a structured method for systematic and integrated occupational safety and health and patient safety management systems (SIOHPS). A process evaluation will be conducted alongside the main study to determine the intervention's specific outcomes and provide transferable guidance to a wider context. The intervention is designed to support both systematic occupational health and patient safety management systems using a Safety II-perspective. The intervention is comprised of several core components, including education to staff, support-functions and management, daily team reflections; as well as audit and feedback.

A stepped wedge cluster-controlled design (SWD) will be used, with workplaces as clusters. The SWD will consist of three steps, with four clusters crossing over from the control to the intervention group at each step. All clusters will start as controls. At least twelve healthcare units with at least thirty employees per workplace from two different regions in Sweden will participate in the intervention. Workplaces that provide round-the-clock care are invited to participate in the study. Exclusion criteria are units with plans to implement any other occupational health and/or patient safety improvement work during the project period. At the individual level, inclusion criteria for employees include at least 50% of full-time work at the workplace.

The SIOHPS project will contribute to the existing theory on safety culture interventions by considering the integration of these areas. The goal is to contribute to a safe environment for both employees and patients.

DETAILED DESCRIPTION:
The increasing and aging populations, changing patient needs and advances in technology present significant challenges to healthcare systems around the world. These challenges are particularly demanding in complex systems associated with high risks, such as the healthcare. In addition to the suffering experienced by patients, preventable adverse events can result in increased loading and costs to the hospitals and challenges in the healthcare work environment. Over the years, reports of poor working conditions in the healthcare sector, characterized by high workload and stress have been raised. Previous studies have shown an association between the work environment and employees´ health, as well as patient outcomes. The evidence unequivocally supports the association between the work environment and patient safety. The negative impact of working conditions on both employee health and the quality of care highlights the potential benefits of integrating these areas. Swedish occupational safety and health legislation and the Patient Safety Act require employers to provide good, safe care and to conduct risk assessments to prevent risks and injuries in the healthcare sector. Consequently, it is proposed that integrated systematic occupational health and patient safety management are crucial in managing the challenges faced by healthcare services today. However, there is a lack of research-based tools and methods to evaluate the impact of integrated systematic occupational health and patient safety management on quality and safety. Moreover, it is essential to evaluate the process of developing, implementing, and utilizing a new tool and method.

The project aims to assess the effectiveness and cost-effectiveness of a structured method for systematic and integrated occupational safety and health and patient safety management systems (SIOHPS). A process evaluation will be conducted alongside the main study to determine the intervention's specific outcomes and provide transferable guidance to a wider context.

The intervention is designed to support both systematic occupational health and patient safety management systems (Safety I) including a Safety II-perspective, i.e. bringing into focus situations where safety is actually present, that is, in everyday work that usually goes well. The content of the intervention is based on the Safer Culture Framework, Swedish regulations related to the field, and current evidence of effective interventions to improve safety culture in healthcare organizations. The intervention is comprised of several core components such as targeted education, daily team reflections and support for systematic management.

First, a two hour education will be conducted for management, health care workers (HCW) involved in patient safety work, safety representatives and intervention facilitators. The education includes information on 1) occupational health and safety as well as patient safety, concepts and systematic management systems, 2) safety culture and psychological safety, 3) demonstration of the content of the intervention including the supporting digital tool and 4) case discussions. All HCW will take part of a short version of the education (approximately 30 minutes) with similar content. The education sessions will be delivered to each cluster close to intervention start. The second core component is a short daily team reflection conducted by HCW at the unit in connection to the end of work shifts. These are standardized to support identification of situations at work related to both Safety I and II perspective for both occupational health and patient safety as well as learning. The facilitator supports the HCW in the process of the daily reflections to maintain adherence and sustainability. The third component includes risk assessment, planning and implementation of appropriate measures, follow-up and feedback, based on information identified in the second component. The steps in this component targets the management and should be conducted in close collaboration with HCW involved in patient safety work and the safety representatives. Participation of HCW in this part is encouraged.

The project is guided by the Medical Research Council (MRC) framework for complex interventions and is coproduced with stakeholders. A program theory guides the evaluation of intervention effectiveness. The study has a hybrid Type I design in which the primary aim is to determine effectiveness of an intervention with the secondary aim to better understand context for implementation and evaluate the process.

A stepped wedge cluster-controlled design (SWD) will be used, with units as clusters. The design is suitable in intervention studies where all clusters could benefit from the intervention. A pragmatic randomization procedure will be used upon assignment of steps for each cluster to assure an equal number of clusters and employees in each step. Consideration will be given to geographically neighboring clusters and collaboration between managers when deciding cluster allocation for each step, aiming to minimize the risk of influencing those in the other steps.

The SWD will consist of three steps, with at least four clusters crossing over from the control to the intervention group at each step. The study begins with a period where all clusters function as controls and then, in multiple steps, transition from the control group to the intervention group. The transition to each new step occurs every four months. At least twelve healthcare units with at least thirty employees per workplace from two different regions in Sweden will participate in the intervention. Workplaces that provide round-the-clock care are invited to participate in the study. Exclusion criteria are units with plans to implement any other occupational health and/or patient safety improvement work during the project period; and units providing pediatric and psychiatric care. At the individual level, inclusion criteria for employees include at least 50% of full-time work at the workplace. All professions are included and encourage to participate in the intervention.

A power calculation has been conducted where the effect has been estimated at the employee level (intervention effect) based on the following parameters: Power 80%, p <0.05, clinically relevant change in the primary outcome is 30%, ICC = 0.01, number of "steps" = three, and an equal number of clusters switch to the intervention group at each occasion. Each cluster is assumed to consist of an average of 30 employees, which means that at least twelve clusters need to be included.

The intervention is utilized by participating units for eight months, but units in the initial steps are encouraged to continue using the intervention until the units in the last step have finished their intervention period.

The intervention effect will be evaluated using the primary outcomes sick leave and quality of care. Secondary outcomes include safety climate, work environment-related factors, employee health, performance and patient safety. Primary outcomes are monitored using registry data. Secondary outcomes are collected using questionnaires which will be sent out to all employees in each cluster and step at baseline, 4 months, and 8 months after intervention start. Primary and secondary analyses are conducted based on intention-to-treat. Complementary per-protocol analyses are carried out for both primary and secondary outcomes. Subgroup analyses are considered if the data allows, for instance, based on units, perceived safety climate, gender, healthcare professions, or risk of ill health.

Different complementary data are collected for the cost-effectiveness evaluation. Direct costs for resource usage in the intervention include, for example, the time spent in each meeting and the number of participating employees, consumable materials, etc. Indirect costs include production losses due to work environment and/or health-related issues, as well as absenteeism. Cost-effectiveness is calculated using a cost-benefit analysis and cost-consequence analysis.

The design of the process evaluation is based on Medical Research Council framework and Moore et als. three core components: implementation (how delivery is achieved and what is delivered), mechanisms of impact (how the intervention creates change), and context (how context influences implementation and outcomes). To more comprehensively assess and manage factors that may affect successful implementation of interventions in various contexts, the Consolidated Framework for Implementation Research (CFIR) has been utilized. Prior to study start information will be collected on contextual factors that may have influenced the implementation process and will be assessed by telephone interviews. The data collection for the process evaluation is carried out concurrently with the implementation of the intervention project and data will be collected over the eight months. It will be assessed by documentation, observation, questionnaires and focus group interviews.

Information will be distributed to managers in the Swedish healthcare system, via contact persons such as central patient safety representatives, HR-representatives and work environment specialists. If expressed interest from these functions, continued establishment within the organization will occur through senior management to first line management. Informed consent from senior management will be collected before further contact will be established with first line managers. Information about the study and what participation entails will be sent to managers by email and followed up with information meetings or equivalent. Included units will receive additional information about the study directed towards HCW at the unit. The research group will give further information about the study at workplace meetings with the possibility for the employees to ask questions and receive additional information. The HCW will be invited to participate in the study via their e-mail addresses at work. Informed consent will be collected in conjunction with the baseline questionnaire is sent out. Participation in the study is voluntarily. All HCW are eligible to participate in the intervention regardless of whether they choose to participate in the research study or not.

ELIGIBILITY:
Inclusion Criteria:

* Individual staff needs to work at least 50% at the workplace
* Workplace provides 24-hour care

Exclusion Criteria:

* Plan to implement another method for conduction daily work environment and/or patient safety work during the project period
* Units providing pediatric and psychiatric care

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Sick leave | 12 months
  Total number of sick leave days after intervention start. Register data.
Quality of care | 12 months
  Readmission rate within 30-days of discharge. Register data.

SECONDARY OUTCOMES:
Job demands | 4, 8 months
  Change in perceived job demands at 4 and 8 months after intervention start. Consists of the domains quantitative demands, work pace and emotional demands. Questionnaire data.
Job resources | 4, 8 months
  Change in perceived job resources at 4 and 8 months after intervention start. Job resources includes local leadership, teamwork climate, horizontal trust, meaningful work, influence at work. Questionnaire data.
Learning environment | 4, 8 months
  Change in perceived learning at 4 and 8 months after intervention start. Questionnaire data.
Safety climate | 4, 8 months
  Change in perceived safety climate at 4 and 8 months after intervention start. Includes both occupational health and safety climate as well as patient safety climate. Questionnaire data.
Work environment | 4, 8 months
  Change in perception of the work environment at 4 and 8 months after intervention start. Questionnaire data.
Work Engagement | 4, 8 months
  Change in work engagement at 4 and 8 months after intervention start. Questionnaire data.
Productivity loss | 4, 8 months
  Change in lost productivity at 4 and 8 months after intervention start. Defined as productivity loss related to work environment- and health-related problems. Questionnaire data.
Health | 4, 8 months
  Change in perceived health status of the employees at 4 and 8 months after intervention start. Health is measured as general health, sleep problems, stress, health- and work environment-related problems, exhaustion. Questionnaire data.
Short-term sick leave | 12 months
  Total number of short-term sick leave days after intervention start. Register data.
Quality of care | 4, 8 months
  Change in perceived quality of care at 4 and 8 months after intervention start. Questionnaire data.
Patient Safety | 4, 8 months
  Change in perceived patient safety at 4 and 8 months after intervention start. Questionnaire data.
Incremental cost effectiveness ratios (ICER): Sick leave and Quality of care | 4 months before first intervention enrollment to 8 months after last intervention enrollment
  Evaluation of cost-effectiveness by using calculated costs related to intervention primary outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Region Dalarna, Falun
  - Region Västmanland, Västerås

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.researchweb.org/is/foultv/project/279396

REFERENCES:
- [Derived] Goras C, Ersson AS, Hellman T, Bjurling-Sjoberg P, Bergstrom G, Sarkadi Kristiansson R, Lohela-Karlsson M. Process Evaluation of a Structured Method for Systematic and Integrated Occupational Safety and Health and Patient Safety Management Systems (SIOHPS): Protocol for a Convergent Parallel Mixed Methods Study. JMIR Res Protoc. 2026 Jan 27;15:e89185. doi: 10.2196/89185. PMID 41592318
- [Derived] Lohela-Karlsson M, Ersson AS, Hellman T, Conden Mellgren E, Bergstrom G, Bjurling-Sjoberg P, Sarkadi Kristiansson R, Goras C. Effectiveness- and cost effectiveness of a structured method for systematic and integrated occupational safety and health and patient safety management systems (SIOHPS) - a study protocol for a pragmatic stepped wedge cluster randomised controlled trial. BMC Health Serv Res. 2025 Oct 22;25(1):1391. doi: 10.1186/s12913-025-13537-4. PMID 41126149